CLINICAL TRIAL: NCT05855902
Title: Art Therapy in an Intensive OCD Program: Client Perception of Value
Brief Title: Art Therapy in an Intensive OCD Program
Status: Enrolling by invitation | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 5341
Record Dates: First submitted 2023-03-27; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-05

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with OCD: Adults with OCD in an intensive treatment program will participate in weekly Art Therapy sessions during their enrollment in the program. Each group is 1.5 hours long. Each participant will be asked to fill out one survey after their first Art Therapy group, and one at the end of the time in the program. Both surveys pertain to their perceptions of the value of Art Therapy within the program.
  Interventions: Behavioral: group art therapy

INTERVENTIONS:
Behavioral: group art therapy — Art therapy will be offered in a weekly 1.5 hour group. Clients are provided a prompt and then asked to express their feelings using art, such as drawing/painting/etc.

SUMMARY:
The Thompson Centre Intensive Treatment program for individuals with severe Obsessive-Compulsive Disorder was launched in 2017.

The program is focused on the principles and use of Exposure and Response Prevention Therapy (ERP) and Cognitive Behavioural Therapy (CBT) in its work with clients, however it also integrates other treatment approaches in its structure, including Dialectical Behavior Therapy, Mindfulness, Acceptance and Commitment Therapy, and Art Therapy. Clients are expected to participate in Art Therapy group in the same way they are expected to participate in all other groups in the program schedule.

Though clients comment informally on the benefits of Art Therapy as experienced in the program, study is needed to better understand and appreciate the role Art Therapy can play in helping clients with OCD to manage and where possible, ameliorate, the burden of their symptoms.

Although Art Therapy has been researched to some degree, in particular its role in alleviating distress associated with various health and mental health conditions, to date there has been no systematic investigation addressing or supporting patients'/clients' perception of the value of Art Therapy by people who live with Obsessive Compulsive Disorder (OCD).

In this study, the investigators are proposing to use information from client surveys regarding their experiences in an Art Therapy group within an intensive OCD treatment program, regarding their experience and opinions about the benefits of Art Therapy within a structured, intensive program for individuals who live with severe OCD. Therefore, this proposed study would be an entirely new contribution both to the fields of Art Therapy and OCD.

The hypothesis of the study is that individuals with severe Obsessive-Compulsive Disorder participating in an intensive CBT/ERP treatment program will report benefits specific to their experience in Art Therapy sessions within the program.

DETAILED DESCRIPTION:
Objective:

To evaluate patients'/clients' perceptions of the value of art therapy as a treatment component in an intensive CBT/ERP program for individuals with severe OCD.

To this end, survey responses will be collected from clients in the program and analyzed to identify key benefits of including Art Therapy as a component of their treatment experience.

Study logistics:

All clients in the Intensive Treatment Program are expected to attend all groups, Art Therapy included.

Clients will be informed by staff at the beginning of the program, and by the PI in the first Art Therapy group attended, about the study and will be requested to fill out questionnaires they will receive.

After the first Art Therapy group they will be asked to fill out and submit the first questionnaire. After their last group in the program they will be asked to fill out a final questionnaire.

Those who have already completed the program have submitted completed questionnaires and the data from this will be analyzed retrospectively. The data has been de-identified.

Those who begin the program in June will also be offered a beginning and closing questionnaire, and written consent will be sought to use this data for the prospective part of the study.

Method:

Clients who participate in weekly Art Therapy group will be given one questionnaire to complete after their first art therapy group, and one to complete after their tenth group/tenth week in the program. The questionnaire will be a revised version of the questionnaire that has been given to the clients for the retrospective study data gathering.

Data Analysis:

Clients in an intensive OCD residential/day treatment program - men and women age 18 and up are given two electronic surveys, one at the beginning of their 10-week treatment experience, asking questions pertaining to their experience of Art Therapy after their first session, and at the end of their time in the program, asking them to reflect on their overall experience of Art Therapy in the program.(surveys attached). A descriptive statistical analysis will be used to analyze study data.

Procedures for confidentiality/anonymity:

Participant information will be stored on REDCAP, a confidential and encrypted platform for data collection and storage. All participants will have identifying numbers that are de-linked from their names. This date is password-protected: only the research team will have access to this information.

ELIGIBILITY:
Inclusion Criteria:

* Must have been accepted into and begun the Intensive Treatment Program for OCD at the Thompson Centre, whether participating as a residential or day treatment participant.

Exclusion Criteria:

* No other patients/clients in the hospital or its outpatient programs will be considered for this study. No-one who is not a patient or client in this program can participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with Obsessive-Compulsive Disorder, enrolled in the Thompson Centre Intensive Treatment Program.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-03-23 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Art Therapy Questionnaire | October 2020 - November 2023
  Acceptability of art therapy as rated by scores on the Art Therapy Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Linda E Chapman, M.C.A.T., Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada